CLINICAL TRIAL: NCT00187460
Title: Enhanced Feedback for Effective Cardiac Treatment (EFFECT)
Brief Title: Study of the Effectiveness of Report Cards on the Quality of Care for Heart Attack and Heart Failure Patients
Acronym: EFFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Dr. Jack V. Tu, PI, Institute for Clinical Evaluative Sciences
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CRT43823
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2005-05

CONDITIONS: Acute Myocardial Infarction; Congestive Heart Failure
Keywords: Acute myocardial infarction; Congestive heart failure; Quality of care; Reperfusion; Report cards; Quality indicators
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Feedback Arm (Active Comparator): Hospital corporations randomized to receive early feedback in the form of a report card
  Interventions: Behavioral: Publicly released hospital cardiac report cards
- Delayed Feedback Arm (Active Comparator): Hospitals randomized to receive delayed feedback in the form of a hospital report cared, 21 months after the early feedback arm.
  Interventions: Behavioral: Publicly released hospital cardiac report cards

INTERVENTIONS:
Behavioral: Publicly released hospital cardiac report cards — Participating hospital corporations were randomized to either early feedback or delayed feedback (21 months later) in the form of publicly released hospital report cards of performance on a set of cardiac process-of-care quality indicators.

SUMMARY:
Randomized cluster trial of cardiac report cards for AMI and CHF. 103 acute care Ontario hospitals/85 hospital corporations participating, randomized to two groups: Group A Early Feedback and Group B Delayed Feedback.

Two phases of retrospective chart review of AMI and CHF separations to assess the impact of the public release of hospital specific performance on a set of Canadian quality indicators.

DETAILED DESCRIPTION:
Study Overview:

The EFFECT Study is one of the largest and most comprehensive initiatives in the world to measure and improve the quality of cardiac care. A randomized trial of cardiac care report cards, the study's objective is to determine whether developing and publishing report cards based on clinical data collected from patient charts leads to greater use of evidence-based therapy at hospitals that receive them.

The three-phase study focuses on acute myocardial infarction (AMI) and congestive heart failure (CHF) and involves 85 hospital corporations (consisting of 103 acute care hospitals) in Ontario. As part of the study design, the hospitals were randomized into two groups: Group A-Early feedback hospitals (44 hospital corporations/53 hospitals) and Group B-Delayed feedback hospitals (41 hospital corporations/50 hospitals).

Phase I A retrospective chart review of hospitalizations from 1999/00 and 2000/01 was conducted in the participating Ontario hospital corporations. Findings from Phase I were documented in two reports:

* Report 1. Report Cards on Group A-Early Feedback Hospitals, released January 2004;
* Report 2. Report Cards on Group B-Delayed Feedback Hospitals, to be released September 2005.

In addition to demographic and treatment information, study data also focus on two sets of quality indicators-one for AMI care and one for CHF care. Canadian Cardiovascular Outcomes Research Team (CCORT) investigators, in conjunction with the Canadian Cardiovascular Society (CCS), formed two expert panels to define Canadian AMI and CHF Quality Indicators. The expert panels' membership included clinical leaders in cardiology, internal medicine, family practice, nursing, pharmacy and epidemiology. The indicators are posted on the CCORT web site (www.ccort.ca) and have been published in the Canadian Journal of Cardiology. The study's Technical Advisory Committee reviewed all of the proposed AMI and CHF quality indicators and recommended a final list of indicators for inclusion in the EFFECT report cards.

Phase II Report Cards for Group A-Early Feedback Hospitals and Group B-Delayed Feedback Hospitals based on a second phase of retrospective chart review of 2004/05 hospitalizations. (Release in 2006/07)

Phase III Final Report-Impact Assessment: A comparison of results/improvement from Phase I to Phase II. (Release in 2006/07)

Sources of Funding The EFFECT study is being funded by the Canadian Institutes of Health Research (CHIR) Interdisciplinary Health Research Team (IHRT) Program and the Heart and Stroke Foundation of Canada, with in kind support from the Institute for Clinical Evaluative Sciences.

Principal Investigators The EFFECT study is being led by Dr. Jack V. Tu, MD, PhD, Senior Scientist, ICES, Canada Research Chair, Health Services Research.

ELIGIBILITY:
Inclusion Criteria:

Hospital: Treat > 30 AMI/CHF cases/patients per year in Ontario

Patient:

* AMI Most responsible diagnosis of acute myocardial infarction(ICD-9 code 410)
* CHF Most responsible diagnosis of heart failure(ICD-9 code 428)

Exclusion Criteria:

Patient

* AMI Not admitted to an acute care hospital
* AMI Age < 20 or > 105 years
* AMI Invalid health card number
* AMI Admitted to non-cardiac surgical service
* AMI Transferred from another acute care facility
* AMI coded as an in-hospital complication
* AMI admission within the past year
* CHF Not admitted to an acute care hospital
* CHF Age < 20 or > 105 years
* CHF Invalid health card number
* CHF Admitted to surgical service
* CHF Transferred from another acute care facility
* CHF coded as an in-hospital complication
* CHF admission within the past three years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46000 (Actual)
Dates: Start 2001-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
EFFECT AMI Composite Quality Indicator in the year after report cards published | April 1, 2004 - March 31, 2005
EFFECT CHF Composite Quality Indicator in the year after report cards published | April 1, 2004 - March 31, 2005

SECONDARY OUTCOMES:
CCORT/CCS Individual AMI Quality Indicators in the year after report cards published | April 1, 2004 - March 31, 2005
CCORT/CCS Individual CHF Quality Indicators in the year after report cards published | April 1, 2004 - March 31, 2005

CONTACTS AND LOCATIONS:
Overall Officials: Jack V Tu, MD PhD FRCPC, Principal Investigator — Institute for Clinical Evaluative Studies, Sunnybrook & Women's College Health Sciences Centre, University of Toronto
Locations (1):
- Institute for Clinical Evaluative Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Result] Tu JV, Donovan LR, Lee DS, Austin PC, Ko DT, Wang JT, Newman AM. Quality of Cardiac Care in Ontario. ICES, Toronto, Ontario, 2004
- [Result] Jackevicius CA, Alter D, Cox J, Daly P, Goodman S, Filate W, Newman A, Tu JV; Canadian Cardiovascular Outcomes Research Team. Acute treatment of myocardial infarction in Canada 1999-2002. Can J Cardiol. 2005 Feb;21(2):145-52. PMID 15729413
- [Result] Lee DS, Austin PC, Rouleau JL, Liu PP, Naimark D, Tu JV. Predicting mortality among patients hospitalized for heart failure: derivation and validation of a clinical model. JAMA. 2003 Nov 19;290(19):2581-7. doi: 10.1001/jama.290.19.2581. PMID 14625335
- [Result] Tu JV, Donovan LR, Lee DS, Wang JT, Austin PC, Alter DA, Ko DT. Effectiveness of public report cards for improving the quality of cardiac care: the EFFECT study: a randomized trial. JAMA. 2009 Dec 2;302(21):2330-7. doi: 10.1001/jama.2009.1731. Epub 2009 Nov 18. PMID 19923205
- See also: Related Info — http://www.ccort.ca/EFFECTStudy/tabid/64/Default.aspx